CLINICAL TRIAL: NCT00327665
Title: A Phase I/II, Randomized, Observer Blinded Study to Evaluate and Compare the Safety, Reactogenicity and Immunogenicity of GlaxoSmithKline Biologicals' Investigational Pneumococcal Vaccine Formulations Versus a Licensed Non-GlaxoSmithKline Biologicals' Vaccine and GlaxoSmithKline Biologicals' Aluminum-based 10-valent Pneumococcal Conjugate Vaccine, in Healthy Elderly Subjects
Brief Title: Study to Evaluate the Safety and Immunogenicity of an Investigational Pneumococcal Vaccine in the Elderly Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 106068; 106072 (Other: GSK); NCT00328003 (obsolete NCT alias)
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Infections, Streptococcal
Keywords: pneumonia; pneumococcal vaccine; elderly subjects; invasive pneumococcal diseases; Prophylaxis
MeSH Terms: conditions — Streptococcal Infections; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (5):
- Group A (Experimental)
  Interventions: Biological: 11-valent pneumococcal vaccine GSK513026
- Group B (Experimental)
  Interventions: Biological: 11-valent pneumococcal vaccine GSK513026
- Group C (Experimental)
  Interventions: Biological: 11-valent pneumococcal vaccine GSK513026
- Group D (Active Comparator)
  Interventions: Biological: Pneumo 23™; Biological: Placebo
- Group E (Active Comparator)
  Interventions: Biological: 10-valent pneumococcal vaccine GSK513026

INTERVENTIONS:
Biological: 11-valent pneumococcal vaccine GSK513026 — Two-dose intramuscular injection. Each group receiving one of the 3 formulations
  Arms: Group A; Group B; Group C
Biological: Pneumo 23™ — Single-dose intramuscular injection.
  Arms: Group D
Biological: Placebo — 1 intramuscular injection.
  Arms: Group D
Biological: 10-valent pneumococcal vaccine GSK513026 — Two-dose intramuscular injection
  Arms: Group E

SUMMARY:
As the licensed pneumococcal vaccine is not always satisfactory in elderly, new investigational pneumococcal vaccines are evaluated in the healthy elderly population. Note: The study consists of the primary phase (106068): vaccination and follow-up and the extension (106072) of the primary phase: 1 year follow-up.

This protocol posting details the procedures of both the primary & extension phase.

DETAILED DESCRIPTION:
No new subjects will be enrolled in the Extension Phase of the study. All outcome measures at Month 12 will only be evaluated in the subjects in the Belgian site.

Upon request, volunteers will receive flu vaccination free of charge. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female between 65 and 85 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.

Exclusion Criteria:

* Previous vaccination against Streptococcus pneumoniae.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory tests.
* Acute disease at the time of enrolment.
* History of documented radiologically confirmed pneumonia within 3 years prior to first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Current or history of Parkinson disease, Alzheimer disease, stroke, dementia or any serious neurologic or mental disorders.
* All malignancies (excluding non-melanic skin cancer) and lymphoproliferative disorders diagnosed or treated actively during the past 5 years.
* Subjects with documented anaemia or iron-deficiency.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 3 months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 2 weeks of the first dose of vaccine(s) with the exception of a Flu vaccine which can be administered at least 1 week preceding the first dose of vaccine(s) or 1 month after the first dose of the vaccine(s).
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of immunoglobulins and/or any blood products within three months preceding the first dose of study vaccine or planned administration during the study period.
* History of administration of an experimental/licensed vaccine containing MPL or QS21.
* History of chronic alcohol consumption and/or drug abuse.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 335 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2007-01-01 (Actual); Study Completion 2007-01-08 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of any solicited local and general signs and symptoms. | during a 7-day follow up period after each vaccine dose.
Occurrence, intensity and relationship to vaccination of unsolicited local and general signs and symptoms | during a 31-day follow up period after each vaccine dose.
Occurrence and relationship to vaccination of all serious adverse events (SAEs). | Throughout the study period.
Post vaccination concentration IgG ≥5 µg/mL and fold increase Post/Pre ≥2 for at least 6 serotypes out of 11 | 1 month after Dose 2 in Groups A, B, C and 1 month after Dose 1 for Group D
Post vaccination concentration and fold increase Post/Pre ≥2 for at least 6 serotypes out of 11, in Groups A through D. | One month after the first vaccine dose.

SECONDARY OUTCOMES:
Haematological and biochemical levels within or outside the normal ranges in all groups. | At Months 0, 1, 3, 4 and 12.
IgG antibody concentrations to vaccine pneumococcal serotypes in all groups. | At Months 0, 1, 3, 4 and 12.
Opsonophagocytic activity titres (OPA) against pneumococcal serotypes in all groups. | At Months 0, 1, 3, 4 and 12
Frequencies of IgG PS-specific plasma cells generated by in vitro cultivated memory B-cells for 4 serotypes in all groups, and for 11 serotypes in 10 subjects per group. | At Months 0, 1, 4 and 12.
Anti-protein D, anti-tetanus and anti-diphtheria toxoids IgG antibody concentrations in Groups A, B, C and E. | At Months 0, 1, 3, 4 and 12.
Frequencies of IgG carrier protein-specific plasma cells generated by in vitro cultivated memory B-cells in a subset of subjects (all subjects minus PS B-cell memory subset) of the Groups A, B, C and E. | At Months 0, 1, 4 and 12.
Freq. of CD4+&CD8+ T cells with antigen-specific IL-2 &/or INFy &/or TNFa &/or CD40L secretion/expression to carrier protein as determined by ICS, in a subset of subjects (all subjects minus PS B-cell memory subset) of the Groups A, B, C and E. | At Months 0, 1, 4 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Ghent, Belgium
- GSK Investigational Site, Pirkkala, Finland
- GSK Investigational Site, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 106068 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/106068?search=study&b''#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 106068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106068 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register